CLINICAL TRIAL: NCT04662333
Title: Adjunctive Benefit of Xenograft Plus a Membrane During Sinus Crestal Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLS001
Record Dates: First submitted 2020-11-29; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Edentulous Jaw
Keywords: Dental implant; Sinus lift; maxillary atrophy; biomaterials
MeSH Terms: conditions — Jaw, Edentulous; Atrophic Maxilla

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crestal sinus lift (Active Comparator): Implant site preparation with detachment of Schneiderian membrane and subsequent implant placement. The corresponding healing abutment is made up of PEEK (poly-ether-ether-ketone)
  Interventions: Procedure: Transcrestal approach for sinus lift
- Crestal sinus lift with adjunctive xenograft (Experimental): Implant site preparation with detachment of Schneiderian membrane. After that, collagen membrane plus xenogenic bone substitute will be placed into the site before implant placement. The corresponding healing abutment is made up of titanium.
  Interventions: Procedure: Transcrestal approach for sinus lift; Procedure: Xenograft application

INTERVENTIONS:
Procedure: Transcrestal approach for sinus lift — After surgical exposure of maxillary alveolar crest, implant site preparation and transcrestal detachment of Schneiderian's membrane will be performed. Thereafter implant will be placed, protruding in the maxillary sinus with its apical part.
Procedure: Xenograft application — Before implant placement, xenogenic collagen membrane and bone granules will be pushed under the Schneiderian's membrane through the surgical site.
  Arms: Crestal sinus lift with adjunctive xenograft

SUMMARY:
Patients in need for implant-supported restoration in maxillary posterior sites with insufficient residual bone height will be randomly allocated to two different arms. Crestal sinus lift with simultaneous implant placement will be performed in both groups.

Control group: crestal sinus lift with no adjunctive biomaterial; Test group: crestal sinus lift associated with xenogenic bone graft and collagen membrane; Six months after implant placement, implants will be loaded with definitive screw-retained prostheses.

Six months later, patients will be recalled for clinical and radiographic assessment.

DETAILED DESCRIPTION:
Patients in need for implant-supported restoration in maxillary posterior sites with bone deficiencies will be randomly allocated to two different arms.

Full-mouth periodontal chart and standardized radiographs will be evaluated at the time of inclusion.

Crestal sinus lift with simultaneous implant placement will be performed in both groups.

Control group: crestal sinus lift with no adjunctive biomaterial; the healing abutment in this group is made up of PEEK (poly-ether-ether-ketone).

Test group: crestal sinus lift associated with xenogenic bone graft and collagen membrane; the healing abutment in this group is made up of titanium;

Resonance frequency analysis will be performed at the time of implant placement and at 1, 3, 6 months of follow-up.

Both healing abutment will be undersized: this characteristic will allow to harvest a 1mm-wide biopsy of the transmucosal tract at the end of the healing phase (6 months).

Six months after implant placement, impression will be taken and implants loaded with definitive screw-retained prostheses.

Six months later, patients will be recalled for clinical and radiographic assessment.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* edentulous in posterior maxilla
* patient in need of sinus augmentation procedure
* residual bone height greater than 3mm

Exclusion Criteria:

* systemic chronic diseases affecting osseointegration
* contraindication for implant therapy
* less than 18 years
* uncontrolled periodontitis
* smoker (more than 10 cig/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Complications rate | 12 months
  amount of complications assessed at patient level

SECONDARY OUTCOMES:
Peri-implant bone stability | 12 months
  the amount (mm) of crestal bone resorption after implant placement assessed through intraoral radiographs
Implant stability quotient | baseline, 1 month, 3 months, 6 months
  implant stability assessed by resonance frequency analysis
Soft tissue inflammation | 6 months
  percentage of peri-implant soft tissue affected by inflamed connective tissue

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, Italy